CLINICAL TRIAL: NCT02526303
Title: Anticoagulation for Non-occlusive Portal Vein Thrombosis in Patients With Liver Cirrhosis: a Single Center Prospective Randomized Controlled Trial
Brief Title: Anticoagulation for Non-occlusive Portal Vein Thrombosis in Patients With Liver Cirrhosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PVT-AT-1
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Liver Cirrhosis; Portal Vein Thrombosis; Anticoagulation
MeSH Terms: conditions — Liver Cirrhosis | interventions — Nadroparin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anticoagulation (Experimental): Drug: Nadroparin Calcium and Warfarin Patients will take warfarin started at a dose of 2.5mg/d and with titration of dose to maintain a target INR of 2-3,along with Nadroparin Calcium 85IU／kg，subcutaneous, q12h,for the first 5 days at least.
  Interventions: Drug: Nadroparin Calcium and Warfarin
- Non-anticoaglated (No Intervention): No anticoagulatoin or other treatment for PVT will be used in this group of patients.

INTERVENTIONS:
Drug: Nadroparin Calcium and Warfarin — Warfarin (with nadroparin calcium at the first 5 days at least) until recanalization or 1 year
  Arms: Anticoagulation

SUMMARY:
The purpose of this study is to determine the safety and efficacy of anticoagulation in the treatment of non-occlusive portal vein thrombosis in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Portal vein thrombosis is a common complication of liver cirrhosis, especially at the decompensated or advanced stage. The reported prevalence was 10-25% by ultrasound. The effect of PVT on the natural history of liver cirrhosis is not clear, especially the non-occlusive PVT. According to a recent large prospective study (n=1243), the development of PVT and the progression of liver disease are two separate consequences of a common mechanism. It was hypothesized that the activation of coagulation factors in the cirrhotic liver or the portal venous system is the common mechanism for the progression of liver disease, on the one hand, and the development of PVT on the other. A recent randomized clinical trial has shown that enoxaparin therapy for 48 weeks can prevent disease progression and PVT in patients with Child class B-C cirrhosis. Besides, emerging evidences have shown that 30-50% of patients with cirrhosis and partial PVT can achieve this spontaneous recanalization. So what the role of anticoagulation played in the management of PVT in liver cirrhosis is still contraversal. Anticoagulation therapy was also shown very effective with a high recanalization rate of 42-100%. But this data was mostly derived from retrospective, non-randomized study and no well-designed randomized controlled trial has been conducted to evaluate the safety and efficacy of anticoagulation for non-occlusive PVT.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent was obtained
* liver cirrhosis
* Non-occlusive portal vein thrombosis
* No history of variceal bleeding or receive endoscopy or β-blocker for the prevention of patients with G3 or G2 with red marks within 3 months before enrollment
* No plan for liver transplantation
* Age between 18 and 70
* Child-Pugh score ≤ 11

Exclusion Criteria:

* Acute PVT
* Fibrotic cord of PV
* Isolated splenic vein thrombosis or isolated superior mesenteric vein thrombosis
* Extensive superior mesenteric vein thrombosis involving the distal part
* Known coagulation disorder besides liver cirrhosis
* HCC or other malignant tumor
* Patients with G2 varices with red mark or G3 but did not underwent any preventive endoscopy or β-blockers
* Platelet count < 10×109/L
* Receive contraceptive, anticoagulation or antiplatelet drug
* Receiving thrombolysis treatment
* Receiving TIPS or shunting surgery
* Bleeding tendency
* Recent gastrointestinal bleeding like digestive ulcer or hemorrhagic stroke
* Severe portal hypertension，for example, refractory ascite or acute variceal bleeidng
* Spontaneous bacterial peritonitis
* Severe cardiovascular disorder, endocrine disorder, or mental disease
* Major surgery within 6 months
* History of organ transplantation
* Pregnancy or breast-feeding
* History of HIV
* Poor compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Portal Vein Recanalization as Assessed by Cummulative Rate | 2 year

SECONDARY OUTCOMES:
Number of Participants With Liver Decompensation as Assessed by Cummulative Rate | 2
Number of Participants Who Show Improvement in Child-Pugh score > 2 Points | 2 years
  Child-Pugh Scores range from 5 to 15
Number of Participants Who Show Improvement in MELD Score > 5 points | 2 year
Number of Participants with Improved Stiffness of liver and Spleen as Assessed by Transient Elastography | 2 years
Number of Participants with Recurrence of Thrombotic Events as Assessed by Cummulative Rate | 2 years
Number of Participants Who still Alive at the end of trial as Assessed by Cummulative Rate | 2 years
Relationship between Portal Vein Recanalization and Survival Assessed by Cox's Regression Proportional Hazard Model | 2 years
Number of Participants With Major Bleeding as Assessed by Cummulative Rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, PhD,MD, Principal Investigator — Xijing Hospital of Digestive Diseases, Fourth Military Medical University

REFERENCES:
- [Background] Qi X, Han G, Fan D. Management of portal vein thrombosis in liver cirrhosis. Nat Rev Gastroenterol Hepatol. 2014 Jul;11(7):435-46. doi: 10.1038/nrgastro.2014.36. Epub 2014 Apr 1. PMID 24686266
- [Background] Nery F, Chevret S, Condat B, de Raucourt E, Boudaoud L, Rautou PE, Plessier A, Roulot D, Chaffaut C, Bourcier V, Trinchet JC, Valla DC; Groupe d'Etude et de Traitement du Carcinome Hepatocellulaire. Causes and consequences of portal vein thrombosis in 1,243 patients with cirrhosis: results of a longitudinal study. Hepatology. 2015 Feb;61(2):660-7. doi: 10.1002/hep.27546. Epub 2015 Jan 5. PMID 25284616
- See also: Click here for more information about this study:Management of portal vein thrombosis in liver cirrhosis — http://www.nature.com/nrgastro/journal/v11/n7/full/nrgastro.2014.36.html